CLINICAL TRIAL: NCT05743166
Title: Bariatric Surgery Observation Study Part 2 An Observational Study of Patients Who Underwent Bartiatric Surgery in Public Hospitals in Central Norway 2010-2015.
Brief Title: Bariatric Surgery Observation Study Part 2
Acronym: BAROBS2
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: Helse Nord-Trøndelag HF (Other); Helse Møre og Romsdal HF (Other Government)
Responsible Party: Sponsor
Other Study IDs: StOlavsH
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — JDF11 JDF41 JDF97
  Other Names: Roux-en-Y gastsric bypass; Sleeve gastrectomy

SUMMARY:
The goal of this observational study is to explore the longterm effects of two bariatric surgical procedures by inviting patients from three public hospitals who had Roux-en-Y gastric bypass or Sleeve gastrectomy to a follow-up after10-15 years

The main question[s] it aims to answer are:

* The duration of the surgical method on weight reduction and remission of comorbidities
* Theprevalence of complications and new morbidities after the surgical procedures Participants will be asked be asked to

  * fill inn questionnaires,
  * have a clinical examinition
  * have an interview with nurse and doctor
  * have blood samples taken
  * undergo other investigations

DETAILED DESCRIPTION:
The BAROBS project is a collaberation between three public hospitals in Norway exploring the concequeces ten years or more after undergoing gastric bypass or sleeve gastrectomy for severe obesity.

1400 patients who underwent bariatric surgery at the three hospitals will be invited to a follow up including antrophometric, meassurment of bodily composition by bioimpedance and DXA, blood samples, questionnaires on sosioeconomic topics, symptoms and quality of life, continous glucose monitoring, dental examination, and other clinical evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric surgery at Namsos Hospital, St. Olavs hospital or Ålesund Hospital from 01.01.2010 to 31.12.2015

Exclusion Criteria:

* Not able to consent for participation
* Includable participants not longer living in Norway

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1400 patients who had baratric surgery at three public hospitals in Central Norway from 2010 to 2015 are invited to a follow up in 2023-2025
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-28 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Long-term weight loss | 10-15 years after surgery
  Total weight loss after bariatric surgery

SECONDARY OUTCOMES:
Remission of comorbidities after bariatric surgery | 10-15 years after surgery
  Remission of Type 2 Diabetes Mellitus, Hypertension and Sleep Apnoe
Quality of life after bariatric surgery | 10-15 years after surgery
  Health related quality of life, SF -36

CONTACTS AND LOCATIONS:
Overall Officials: Jorunn Sandvik, PhD, Principal Investigator — St. Olavs Hospital
Locations (3):
- Norway (3):
  - Helse Møre og Romsdal, Ålesund
  - Helse Nord-Trondelag, Namsos
  - St. Olavs Univeristy Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No